CLINICAL TRIAL: NCT04625738
Title: Efficacy of Infusions of Mesenchymal Stem Cells From Wharton Jelly in the Moderate to Severe SARS-Cov-2 Related Acute Respiratory Distress Syndrome (COVID-19): A Phase IIa Double-blind Randomized Controlled Trial
Brief Title: Efficacy of Infusions of MSC From Wharton Jelly in the SARS-Cov-2 (COVID-19) Related Acute Respiratory Distress Syndrome
Acronym: MSC-COVID19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, POCHON Cécile, Coordinator, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-002772-12
Record Dates: First submitted 2020-11-04; First posted 2020-11-12 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: COVID19 ARDS
Keywords: COVID; ARDS; MSC; mesenchymal stem cells; Wharton's Jelly; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Phase IIa double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MSC Arm (Experimental): Ex vivo expanded Wharton's Jelly derived mesenchymal stem cells will be infused at day 0, day 3 and day 5 (+/- 1 day), in patients with moderate to severe ARDS with a mechanical ventilation.
  day 0: 1.10^6 MSC/kg day 3: 0.5. 10^6 MSC/kg day 5: 0.5 . 10^6 MSC/kg
  Interventions: Biological: Ex vivo expanded Wharton's Jelly Mesenchymal Stem Cells
- Placebo Arm (Placebo Comparator): Only the vehicle solution, without MSCs, containing albumin 4% , NaCl 0,9% and ACD will be injected to patients at day 0, 3 and 5 (+/-1 day).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ex vivo expanded Wharton's Jelly Mesenchymal Stem Cells — Ex vivo expanded Wharton's Jelly derived mesenchymal stem cells will be infused at day 0, day 3 and day 5 (+/- 1 day), in patients with moderate to severe ARDS with a mechanical ventilation.
  day 0: 1.10^6 MSC/kg day 3: 0.5. 10^6 MSC/kg day 5: 0.5 . 10^6 MSC/kg
  Arms: MSC Arm
Biological: Placebo — Only the vehicle solution, without MSCs, containing albumin 4% , NaCl 0,9% and ACD will be injected to patients at day 0, 3 and 5 (+/-1 day).
  Arms: Placebo Arm

SUMMARY:
Mesenchymal stem cells (MSCs) are of potential help in acute respiratory distress syndrome (ARDS), due to their anti-inflammatory properties.

The investigators will analyze the effect of 3 iterative infusions of ex vivo expanded Wharton's Jelly MSCs (total dose 2.10^6/kg) in patients with ARDS due to COVID19, who require mechanical ventilation.

DETAILED DESCRIPTION:
This study is designed to analyze the impact of Wharton's Jelly Mesenchymal Stem Cells on moderate to severe ARDS due to COVID19 in adult patients who require mechanical ventilation. It is a Phase IIa double-blind randomized controlled trial.

30 patients are planned.

Patients will be randomized and will receive, with the conventional treatment recommended to treat ARDS:

* Either Wharton's Jelly MSCs in a solution of albumin 4% (40% of final volume), NaCl 0,9% (50% of the final volume) et ACD formule A (10% of the final volume) . Treatment will be administered intravenously during 10 minutes following that scheme:

  * Day 0 (or 1): 1. 10^6 MSC/kg (maximum 80.10^6 MSC)
  * Day 3 (or 4): 0.5 . 10^6 MSC/kg (maximum 40. 10^6 MSC)
  * Day 5 (or 6): 0.5 . 10^6 MSC/kg (maximum 40. 10^6 MSC) An interval of 2 days will be respected between 2 infusions.
* Either a placebo, which contains the same solution of albumin, NaCl 0.9% and ACD without cells. The volume will be of 75 ml, infused in 10 minutes.

The main objective is to investigate efficacy of WJ-MSCs, compared to a placebo, on respiratory function evolution during the first 14 days of study treatment in patients with SARS-CoV-2 related moderate to severe ARDS.

Secondary objectives are to assess the effect of WJ-MSC, compared to placebo, in patients with SARS-CoV-2 related moderate to severe ARDS, on:

1. the duration of invasive mechanical ventilation during the hospital stay and maximum for 28 days
2. the evolution of organ failures during the hospital stay and maximum for 28 days
3. the duration of stay in intensive care unit, the mortality during intensive care unit, during hospitalization, on D28 and D90, and the respiratory morbidity.
4. the evolution of viral load between D0 and D28
5. the immediate or delayed tolerance following the WJ-MSCs injection

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman 18 years of age or older
2. Patient with a biologically confirmed SARS-CoV-2 infection (by positive RT-PCR on a nasopharyngeal sample or any other sample)
3. Patient with moderate to severe ARDS according to the BERLIN definition defined by a PaO2 / FiO2 ratio <200 and with endotracheal intubation and under invasive mechanical ventilation
4. Patient hospitalized in the intensive care unit
5. Provision of a written informed consent to participate to the study or for whom the consent of a family member or support person has been obtained (if the patient is unable to give consent) or inclusion in an immediate vital emergency if applicable
6. Any woman of childbearing age with a negative Beta HCG test
7. Social Security affiliation

Exclusion Criteria:

1. Patient under invasive mechanical ventilation for more than 48 hours
2. Patient with a chronic respiratory disease under oxygen therapy
3. Patients with a history of Class III or IV pulmonary arterial hypertension (WHO classification)
4. Patients under ECMO
5. Immunosuppressive therapy (including corticosteroid therapy> 20 mg prednisolone)
6. Active solid tumor or in remission for less than 2 years, malignant hematological disease, asplenia
7. Patient who has received a hematopoietic stem transplantation or an organ transplant
8. Therapeutic limitations like progression to expected death within 24 hours (according to the opinion of the medical team)
9. Hypersensitivity to albumin or to any of the excipients (caprylic acid or sodium caprylate)
10. Patient included in another ongoing interventional therapeutic trial
11. Pregnant woman, parturient, nursing mother
12. Minor (not emancipated)
13. Person without liberty by judiciary or administrative decision
14. Person undergoing psychiatric care under Articles L. 3212-1 and L. 3213-1 which do not fall under the provisions of Article L. 1121-8 (hospitalization without consent).
15. Adult over 18 who are under a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
PaO2 / FiO2 ratio | day 10
  The primary endpoint is the percentage of patients with a PaO2/FiO2 ratio > 200 at D10 of treatment with MSC-GW or placebo.

SECONDARY OUTCOMES:
respiratory function evolution | between Day 0 (or Day 1) and Day 14 of treatment
  The evolution of the PaO2/FiO2 ratio between Day 0 (or Day 1) and Day 14 of treatment with MSC-GW or placebo is a secondary endpoint.
respiratory assistance | between day 0 (or 1) and day 28 (or last day of hospitalization if before day 28)
  The effect of WJ-MSC on respiratory assistance is evaluated by the proportion of days without invasive respiratory assistance during the hospital stay and maximum on Day 28 (number of days without invasive respiratory assistance / number of hospital days fixed at day 28)
organ failures 1 | Day 0 to day 14
  Difference in sequential organ failure assessment score (SOFA score), grading 0 (best) to 4 (worst), between Day 5-Day 0 and D14-Day 0
organ failures 2 | day 0 to day 28
  number of days without extra-renal treatment / number of hospital days fixed at day 28
organ failures 3 | day 0 to day 28
  number of days without vasopressor support
duration of intensive care | day 0 to 90
  The duration of stay in intensive care unit
Cause of death | day 0 to 90
  Cause of death during the stay in intensive care unit and during the hospital stay, on Day 28 and Day 90
respiratory morbidity (TDM, functional respiratory measures) | day 90
  respiratory morbidity on Day 90
viral load | day 0 to day 28 (or last day of hospitalization if before day 28)
  The evolution of the viral load is evaluated by RT PCR SARS-Cov-2 monitoring on a nasopharyngeal swab (or any other sample) at diagnosis, at Day 7, Day 14, Day 21, Day 28 or on the last day of hospitalisation
Anti-HLA antibody rate | day 0 to day 90
  - The anti-HLA antibody rate measured on Day 0 (before initiating treatment), on Day 28 and on Day 90
immediate hypersensitivity reactions | day 0, day 3, day 5 (+/- 1day)
  The occurrence of immediate hypersensitivity reactions (chills, hyperthermia associated with hypotension) within 4 to 6 hours of the WJ MSC or placebo infusion.
thromboembolic adverse events 1 | day 0 to day 14
  The thromboembolic risks monitored biologically by routinely daily monitoring of hemostasis (TP, TCA, Fibrinogen, D-dimers)
thromboembolic adverse events 2 | day 0 to day 14
  daily monitoring of transthoracic echocardiography
infectious adverse events | day 0 to day 14
  blood cultures in case of T° > 38,5°C

CONTACTS AND LOCATIONS:
Overall Officials: Antoine KIMMOUN, MD, PhD, Principal Investigator — Central Hospital, Nancy, France; Sébastien GIBOT, MD, PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Nancy University Hospital, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pochon C, Laroye C, Kimmoun A, Reppel L, Dhuyser A, Rousseau H, Gauthier M, Petitpain N, Chabot JF, Valentin S, de Carvalho Bittencourt M, Peres M, Aarnink A, Decot V, Bensoussan D, Gibot S. Efficacy of Wharton Jelly Mesenchymal Stromal Cells infusions in moderate to severe SARS-Cov-2 related acute respiratory distress syndrome: a phase 2a double-blind randomized controlled trial. Front Med (Lausanne). 2023 Aug 29;10:1224865. doi: 10.3389/fmed.2023.1224865. eCollection 2023. PMID 37706025